CLINICAL TRIAL: NCT05426772
Title: Investigation of the Effect of Kinesiotape Applied With Exercise on Muscle Oxygenation With Moxy Muscle Oxygen Monitor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Fatma Nur YILMAZ, Assist. Prof., Bandırma Onyedi Eylül University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-60
Record Dates: First submitted 2022-06-02; First posted 2022-06-22 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Healthy; Sedentary
Keywords: muscle oxygen; kinesio taping; near infrared spectroscopy; exercise
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy sedentary people (Other): Muscle oxygenation and vital signs will be measured before, during, and after of 20 minutes aerobic exercise in an environment where suitable conditions are provided. After 3 days, kinesio taping will be added to the same program and the measurements will be repeated.
  Interventions: Other: exercise and kinesiotaping

INTERVENTIONS:
Other: exercise and kinesiotaping — Exercise: Aerobic exercise will be performed on the treadmill for 20 minutes with a maximum heart rate of 55%-65% and a perceived exertion of less than 3. The Moxy muscle oxygen monitor will take measurements over the quadriceps femoris muscle at this time.
  Kinesiotaping: After 3 days, the same participants will be called for kinesiotaping application. The application will be applied to the quadriceps femoris muscle with the facilitation technique by a physiotherapist who has a kinesio taping training certificate.

SUMMARY:
Kinesio taping (KT) is an elastic adhesive tape with physiological effects, often used in rehabilitation and sports medicine. KT, which can stay in the body for 3 to 5 days, exerts a pulling force on the skin thanks to its wave-like structure and elasticity, and increases the gap between the subcutaneous soft tissue and fascia with its lifting effect. In this way, it reduces the superficial pressure and causes an increase in lymph circulation. In addition, with the effect it creates on the muscles, it allows maximum contraction and relaxation of the muscle and creates positive effects on the deep lymphatics. Another effective approach to increase blood circulation is exercise. Exercise, which is known to have many benefits, has been shown to increase both systemic circulation and muscle blood flow. There are findings in the literature that KT can increase the effectiveness of exercise, but it has been stated that this issue is not clear and more studies are needed. In order to evaluate the effects of KT on increasing the effectiveness of exercise and on circulation, the oxygen saturation of the muscle in the application area can be measured. As a matter of fact, "Moxy muscle oxygen monitor" has been used in the literature, which measures regional oxygen saturation (SmO2) and total hemoglobin (THb) in capillaries under the muscle. The Moxy muscle oxygen monitor is a lightweight (42 g) and small (dimensions: 61 × 44 × 21 mm) device that measures regional blood flow and oxygenation by placing it on the skin non-invasively with near-infrared spectroscopy (NIRS). Its validity in measuring muscle oxygenation was vigorous or fairly good, and its reliability was found to be moderate to high in low-intensity exercises (SROC: r = 0.842-0.993, ICC: r = 0.773-0.992, p < .01). It is thought that the application of KT, which is known to increase lymphatic and venous circulation, together with exercise will increase the amount of oxygen in the muscles. To the best of our knowledge in the literature, no study has been found in which this effect of KT is presented objectively. For this reason, it is aimed to examine muscle oxygenation with the Moxy muscle oxygen monitor, which provides objective data on KT applied with exercise.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being between the ages of 18-40
* Being sedentary (<600 MET-min/week according to the International Physical Activity Questionnaire Short Form)
* BMI <30kg/cm2
* Subcutaneous fat thickness <12mm

Exclusion Criteria:

* Having an open wound or infection in the application area
* Having a chronic illness
* Being pregnant
* Having a psychological disorder
* Having a lower extremity injury in the last 6 months
* Having had any surgical operation involving the lower extremity in the last 6 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Moxy Muscle Oxygen Monitor | Baseline
  The Moxy muscle oxygen monitor is a lightweight (42 g) and small (dimensions: 61 × 44 × 21 mm) device that measures regional blood flow and oxygenation by placing it on the skin non-invasively with near infrared spectroscopy (NIRS). The device, which has data collection and telemetric features, also allows O2 measurement in non-laboratory environments and field-based research. Compared to other NIRS devices, the Moxy muscle oxygen monitor has been shown to be a valid and reliable device for muscle oxygenation. Its validity in measuring muscle oxygenation was strong or very good, and its reliability was found to be moderate to high in low-intensity exercises (SROC: r = 0.842-0.993, ICC: r = 0.773-0.992, p < .01). It has been reported that as exercise intensity increases, its reliability changes inversely.
Moxy Muscle Oxygen Monitor | fourth day
  The Moxy muscle oxygen monitor is a lightweight (42 g) and small (dimensions: 61 × 44 × 21 mm) device that measures regional blood flow and oxygenation by placing it on the skin non-invasively with near infrared spectroscopy (NIRS). The device, which has data collection and telemetric features, also allows O2 measurement in non-laboratory environments and field-based research. Compared to other NIRS devices, the Moxy muscle oxygen monitor has been shown to be a valid and reliable device for muscle oxygenation. Its validity in measuring muscle oxygenation was strong or very good, and its reliability was found to be moderate to high in low-intensity exercises (SROC: r = 0.842-0.993, ICC: r = 0.773-0.992, p < .01). It has been reported that as exercise intensity increases, its reliability changes inversely.

SECONDARY OUTCOMES:
heart rate | Baseline
  heart rate will be evaluated with pulse oximetry
heart rate | fourth day
  heart rate will be evaluated with pulse oximetry

OTHER OUTCOMES:
respiratory frequency | Baseline
  respiratory frequency will be evaluated with pulse oximetry
respiratory frequency | fourth day
  respiratory frequency will be evaluated with pulse oximetry
O2 saturation | Baseline
  O2 saturation will be evaluated with pulse oximetry
O2 saturation | fourth day
  O2 saturation will be evaluated with pulse oximetry
blood pressure | Baseline
  blood pressure will be evaluated with sphygmomanometer. Systolic and diastolic pressures will be assessed.
blood pressure | fourth day
  blood pressure will be evaluated with sphygmomanometer. Systolic and diastolic pressures will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylül University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Balıkesir, Bandırma, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No